CLINICAL TRIAL: NCT07180836
Title: Prevalence and Hematological Characteristics of Hemoglobinopathies: A Cross-Sectional Study From a Tertiary Care Hospital
Brief Title: Prevalence and Hematological Characteristics of Hemoglobinopathies
Status: Completed | Type: Observational
Sponsor: Bacha Khan Medical College (Other)
Responsible Party: Principal Investigator, Malik Shayan Ali Khan, Doctor (Principal Investigator), Bacha Khan Medical College
Other Study IDs: Ref no. 499/BKMC
Record Dates: First submitted 2025-08-30; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Hemoglobinopathies
Keywords: Hemoglobinopathies; Thalassemia; Sickle cell disease
MeSH Terms: conditions — Hemoglobinopathies; Thalassemia; Anemia, Sickle Cell | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Hemoglobinopathies in Mardan and Surrounding Districts: This cohort includes patients diagnosed with various hemoglobinopathies in Mardan and neighboring districts of Khyber Pakhtunkhwa, Pakistan. Participants were assessed for prevalence and hematological characteristics, including complete blood count parameters and disease-specific findings. No intervention was applied; this is an observational, cross-sectional study focused on identifying distribution patterns and hematological profiles of hemoglobinopathies in the study population
  Interventions: Other: No Intervention (Observational Study)

INTERVENTIONS:
Other: No Intervention (Observational Study) — This is an observational, cross-sectional study. Patients with suspected or confirmed hemoglobinopathies were evaluated for prevalence and hematological characteristics using laboratory investigations, without any experimental treatment or therapeutic intervention applied.

SUMMARY:
This study aimed to determine the prevalence and hematological characteristics of hemoglobinopathies in Mardan and surrounding districts of Khyber Pakhtunkhwa (KPK), Pakistan. A descriptive cross-sectional design was conducted at Mardan Medical Complex from January 2021 to January 2023. Blood samples were analyzed using High Performance Liquid Chromatography (HPLC) on the Bio-Rad D-10 analyzer, with complete blood counts performed using Sysmex XN1000. A total of 839 participants were enrolled in this study. The study highlights differences in hematological parameters across hemoglobinopathy types and provides region-specific data to inform public health interventions and screening programs.

DETAILED DESCRIPTION:
Hemoglobinopathies are among the most common inherited disorders worldwide, caused by mutations in globin genes affecting hemoglobin synthesis, structure, and function. They are highly prevalent in South Asia, particularly in Pakistan, where beta-thalassemia is the most frequent single-gene disorder. Despite this, there is limited epidemiological data from Khyber Pakhtunkhwa (KPK), especially in Mardan, where consanguineous marriages are common and contribute to disease burden.

This descriptive cross-sectional study was conducted over a two-year period (January 2021 to January 2023) at the hematology department of Mardan Medical Complex, Pakistan. All patients referred for hemoglobinopathy testing were included. Blood samples (3 mL EDTA) were collected and analyzed for complete blood counts (hemoglobin, RBC count, hematocrit, MCV, MCH, MCHC) using Sysmex XN1000, and hemoglobin variants were identified using High Performance Liquid Chromatography (Bio-Rad D-10 analyzer). A sickling test was performed in cases with abnormal S-window chromatogram findings.

A total of 839 participants were analyzed. Geographic distribution was showed for patients from different nearby regions .

This study provides the first comprehensive regional overview of hemoglobinopathies in Mardan, KPK. The findings of our study will emphasize the need for early detection, genetic counseling, and preventive public health strategies, particularly in communities with high rates of consanguinity. These results might support the development of targeted screening and awareness programs to reduce the burden of hemoglobinopathies in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the Hematology Department of Mardan Medical Complex for hemoglobinopathy testing between Jan 2021 - Jan 2023.
* Patients of either sex.
* Patients who underwent high-performance liquid chromatography (HPLC) and complete blood count (CBC) analysis.

Exclusion Criteria:

* Patients with incomplete or missing laboratory data (CBC or HPLC).
* Patients in whom hemoglobinopathy diagnosis could not be confirmed.
* Cases of anemia due to non-hemoglobinopathy causes (e.g., nutritional anemia, chronic disease).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consisted of patients referred for hemoglobinopathy testing to the Hematology Department, Mardan Medical Complex, Mardan, Khyber Pakhtunkhwa, Pakistan, over a period of two years (January 2021 to January 2023). A total of 839 participants were included in the analysis. These patients were of varying ages (mean age: 10.25 ± 4.87 years), with 55.89% male and 43.87% female, and represented different districts including Mardan, Charsadda, Dir, Buner, and Swabi, with the majority from Mardan (86.41%).
Sampling Method: Non-Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hemoglobinopathies. | At the time of diagnosis / Single assessment at enrollment
  Number of patients diagnosed with each hemoglobinopathy type (e.g., β-thalassemia trait, sickle cell disease, HbE).

SECONDARY OUTCOMES:
Demographic Distribution of Hemoglobinopathies by Age, Gender, and Geographic Area | At the time of diagnosis / Single assessment at enrollment
  The study analyzes the demographic characteristics of patients diagnosed with hemoglobinopathies, including distribution by age groups, gender, and geographic location (Mardan and surrounding districts). This outcome helps to identify patterns of disease occurrence and risk groups within the population. Data are derived from patient records and laboratory-confirmed cases.

CONTACTS AND LOCATIONS:
Overall Officials: Malik Shayan Ali Khan, MBBS, Principal Investigator — Bacha Khan Medical College, Mardan.
Locations (1):
- Mardan Medical Comlex, Mardan, Mardan, KPK, Pakistan